CLINICAL TRIAL: NCT02964026
Title: Retrospective Analysis of Clinical Outcomes Associated With Use of the Pulmonary Artery Catheter (PAC) in Cardiac Surgery Patients Within the Cerner HealthFacts Database
Brief Title: Study of Clinical Outcomes Associated With the Pulmonary Artery Catheter (PAC) in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Andrew Shaw, Professor and Executive Vice Chair Department of Anesthesiology Executive Medical Director, Perioperative Services, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 161377
Record Dates: First submitted 2016-10-18; First posted 2016-11-15 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Thoracic Surgery; Cardiac Surgery; Heart Surgery; Heart Transplant
Keywords: pulmonary artery catheter; Swan-Ganz catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary artery catheter (PAC): Patients received a PAC for monitoring purposes
  Interventions: Device: pulmonary artery catheter
- No pulmonary artery catheter (PAC): Patients did not receive a PAC for monitoring purposes

INTERVENTIONS:
Device: pulmonary artery catheter — PAC must be placed between the day of admission and the day following a qualifying cardiac surgery
  Other Names: Swan-Ganz catheter
  Groups: Pulmonary artery catheter (PAC)

SUMMARY:
The primary objective for this retrospective Electronic Health Record (EHR) analysis is to evaluate the clinical outcomes associated with the utilization of a pulmonary artery catheter (PAC), for monitoring purposes, within patients undergoing cardiac surgeries (isolated coronary artery bypass graft [CABG], valve, aortic surgery, multi-procedures, other complex nonvalvular procedures and heart transplants). The study will be conducted using prospectively collected hospital inpatient data over a duration of over 5 years (Jan. 1, 2010 - June 30, 2015) using a large US electronic health database (Cerner HealthFacts; Kansas City, MO).

DETAILED DESCRIPTION:
A retrospective study will be conducted using prospectively collected hospital inpatient data over a duration of over 5 years (Jan. 1, 2010 - June 30, 2015) using a large US electronic health database (Cerner HealthFacts; Kansas City, MO). Patients who underwent a qualifying cardiac surgery (verified through use of selected valid International Classification of Diseases-9 procedure codes and/or Current Procedural Terminology [CPT] codes) will be included. Each patient's cohort designation will be defined based upon whether he/she did or did not receive a pulmonary artery catheter (PAC) for monitoring purposes. Propensity scores, which take into account patient and hospital demographics, patient comorbidities, surgical type (isolated coronary artery bypass graft [CABG], valve, aortic surgery, multi-procedures, other complex nonvalvular procedures and heart transplants), and pre-operative condition (via an adapted EuroSCORE II) will be utilized to "match" patients who received a PAC for monitoring purposes with those who did not, to form a matched study cohort. Clinical outcomes will be monitored through index visit discharge and up to 90 days post index visit discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoes a qualifying cardiac surgery between Jan 1, 2010 and January 1, 2015. If multiple qualifying surgeries are present, the first in database will be utilized
* Inpatient with a LOS of at least 48 hours
* Treated arm receives a PAC for monitoring purposes within admission date and qualifying cardiac surgical day plus one via specified ICD-9 or CPT-4 codes, or EHR recorded PAC readings

Exclusion Criteria:

* Cardiac surgery patients with age <18 years on index procedure date
* Non-treated arm derived from an institution which does not have database documented use of ICD-9 or CPT-4 PAC placement codes for monitoring purposes [Lessens the likelihood that the untreated arm is indeed treated by ensuring that the patient would likely be coded if he/she had a PAC in place for monitoring purposes]
* Patient record must have the demographics populated of age, gender, and race. ICD-9 diagnosis and procedure codes must be present in record for index visit, as well as medications administered over index visit
* Patient must be treated at a hospital which performs a minimum of 100 qualifying cardiac procedures per year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing an isolated CABG, isolated valve, aortic procedure, complex nonvalvular procedures, multi-procedures or a heart transplant who receives or does not receive a pulmonary artery catheter (PAC) for monitoring purposes
Sampling Method: Probability Sample
Enrollment: 6844 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Hospital mortality during index visit | Admission through up to 180 days (hospital discharge)
Hospital length-of-stay (LOS) | Admission through up to 180 days (hospital discharge)
  Index hospital visit LOS
Hospital readmission | Through 30 days
  Rate of hospital readmissions
Hospital readmission | Through 60 days
  Rate of hospital readmissions
Hospital readmission | Through 90 days
  Rate of hospital readmissions
Major Adverse Cardiac Events (MACE) | Through 30 days
Major Adverse Cardiac Events (MACE) | Through 60 days
Major Adverse Cardiac Events (MACE) | Through 90 days
Major morbidity composite | Through 30 days
Major morbidity composite | Through 60 days
Major morbidity composite | Through 90 days

SECONDARY OUTCOMES:
New organ failure (cardiovascular, respiratory, coagulation, liver systems, renal) | Day 1 to discharge (up to 180 days)
Requirement for mechanical ventilation | Day 1 to discharge (up to 180 days)
Hemorrhage requiring blood transfusion | Day 1 to discharge (up to 180 days)
Acute kidney injury (KDIGO staging) | Day 1 to day 10
Infectious complications | Day 1 to discharge (up to 180 days)
Gastrointestinal complication (hepatic) | Day 1 to discharge (up to 180 days)
Respiratory failure | Day 1 to discharge (up to 180 days)
Sequential Organ Failure Assessment (SOFA) scores | Day 1 to discharge (up to 180 days)
Neurologic complication | Day 1 to discharge (up to 180 days)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Shaw, MB, FRCA, FFICM, FCCM, Principal Investigator — Vanderbilt University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw AD, Mythen MG, Shook D, Hayashida DK, Zhang X, Skaar JR, Iyengar SS, Munson SH. Pulmonary artery catheter use in adult patients undergoing cardiac surgery: a retrospective, cohort study. Perioper Med (Lond). 2018 Oct 25;7:24. doi: 10.1186/s13741-018-0103-x. eCollection 2018. PMID 30386591